CLINICAL TRIAL: NCT05355688
Title: Prospective, Single-centre Post-Market Clinical Follow-up (PMCF) Study to Evaluate Safety and Performance of the DUO Venous Stent
Brief Title: Post-Market Clinical Follow-up (PMCF) Study to Evaluate Safety and Performance of the DUO Venous Stent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Arnsberg (Other)
Responsible Party: Sponsor
Other Study IDs: ASL202101
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Deep Venous Obstructions
Keywords: Venous stent system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study is to evaluate performance and safety of the DUO Venous Stent for the treatment of obstructions of the iliac vein.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide inform consent
2. Patients must be ≥ 18 years of age at the time of consent
3. Estimated life expectancy ≥ 12 months.
4. Body mass index (BMI) <35
5. Patients to whom the DUO Venous Stent can be implanted according to the IFU (this includes acute iliac deep vein thrombosis (DVT), post-thrombotic syndrome, non-thrombotic iliac vein compression (e.g. May-Thurner), non-thrombotic iliac vein compression (e.g. compression from ecstatic or tortuous iliac arteries))
6. As per IFU, clinically significant symptomatic venous outflow obstruction in the iliac venous segment, associated by at least one of the following:

   * CEAP score ≥3
   * VCSS pain score ≥2
7. Subject is willing and able to comply with physician's recommendation for compression therapy -

Exclusion Criteria:

1. Presence or history of clinically significant pulmonary emboli within 180 days prior to enrolment.
2. Uncontrolled or active coagulopathy or known, incorrectable bleeding diathesis
3. Prior surgical or endovascular procedure of the target vessel except for catheter-directed or mechanical thrombolysis for DVT within 90 days prior to the index procedure or prior venoplasty
4. Planned surgical or interventional procedures of the target limb (except thrombolysis and/or thrombectomy in preparation for the procedure or vena cava filter placement prior to stent implantation in patients at high risk for pulmonary embolism) within 30 days prior to or 30 days after the index procedure
5. Previous stenting of the target vessel
6. Combination of stents from different manufacturers
7. Participation in another investigational study in which the subject has not completed all primary endpoints or which involves any investigational drug or device that may potentially confound the results of the study
8. Other comorbidities that, in the opinion of the investigator, would preclude the patient from receiving this treatment and/or participating in study-required follow-up assessments
9. Women who are pregnant or lactating
10. Suspected alcohol or drug abuse
11. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with symptomatic obstruction of the iliac vein
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate at month 12 | 12 months
  The primary patency rate is defined as the percentage of stented target lesions with primary treatment success and without the occurrence of thrombosis of the treated lesion or any re-intervention (surgical interventions on the target vessel) to restore or maintain flow within the treated lesion

SECONDARY OUTCOMES:
Primary patency rates | 30 Days, 6 and 24 months
Secondary patency rates | 30 Days, 6, 12 and 24 months
  Percentage of patients with primary treatment success and without occurrence of permanent loss of flow in the treated segment, irrespective of any reintervention
Revised Venous Clinical Severity Score (VCSS) | 30 Days 6, 12 and 24 month
  The score includes 10 clinical parameters (pain, varicose veins, venous edema, skin hyperpigmentation, inflammation, induration, number of ulcers, durations of ulcers, size of ulcers, and compliance with compression therapy). Each item is graded from zero to three depending on severity (None = 0, Mild = 1, Moderate = 2, Severe = 3).
Clinical Etiological Anatomical Pathophysiological Classification score (CEAP) | 30 Days, 6, 12 and 24 months
  The score for the clinical condition of the chronic venous insufficiency (C0 to C6) will be evaluated whereas C0 is representing the best and C6 the worst condition
Villalta score | 30 Days, 6, 12 and 24 month
  The score includes five symptoms (pain, cramps, heaviness, paresthesia, pruritus) and six clinical signs (pretibial edema, skin induration, hyperpigmentation, redness, venous ectasia, pain on calf compression).Each item is graded from zero (not present)to three (severe).
Device or procedure-related adverse events | 30 Days, 6, 12 and 24 month
Serious adverse events | 30 Days, 6, 12 and 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular center of Klinikum Hochsauerland GmbH, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No